CLINICAL TRIAL: NCT01797133
Title: A Comparative Study of ID Fellow-based Pre-authorization VS. Pharmacist-based Pre-authorization in Reducing Antibiotic Consumptions and Hospital Expenditures
Brief Title: A Comparative Study of ID Fellow-based VS. Pharmacist-based Antibiotic Pre-authorization
Acronym: DUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Pinyo Rattanaumpawan, Asssitant Professor, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 647/2555(EC1)
Record Dates: First submitted 2013-02-17; First posted 2013-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: All Hospitalzied Patients; No Specific Conditions Requires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fellow arm (Active Comparator): Patients in this arm will receive the ID fellow-based antibiotic pre-authorization intervention.
  Interventions: Procedure: ID fellow-based antibiotic pre-authorization
- Pharmacist arm (Active Comparator): Patients in this arm will receive the pharmacist-based antibiotic pre-authorization intervention.
  Interventions: Procedure: Pharmacist-based antibiotic pre-authorization

INTERVENTIONS:
Procedure: ID fellow-based antibiotic pre-authorization — All prescriptions of controlled antibiotics (Piperacillin/Tazobactam, Imipenem/Cilastatin, Meropenem and Doripenem) can be freely prescribed for the first 72 hours. After that, the prescription requires approval. Antibiotic preauthorization program will be operated by ID-fellows, under the supervision of ID staffs.
  Arms: Fellow arm
Procedure: Pharmacist-based antibiotic pre-authorization — All prescriptions of controlled antibiotics (Piperacillin/Tazobactam, Imipenem/Cilastatin, Meropenem and Doripenem) can be freely prescribed for the first 72 hours. After that, the prescription requires approval. Antibiotic preauthorization program will be operated by general pharmacists, under the supervision of ID staffs.
  Arms: Pharmacist arm

SUMMARY:
We will conduct a cluster randomized controlled trial to compare two antibiotic pre-authorization strategies (Fellow-based vs. Pharmacist-based). We believe that amount and duration of antibiotic consumption would be lower in the pharmacist group while the clinical outcome would be equivalent between two groups.

DETAILED DESCRIPTION:
Study design: A cluster randomized controlled trial Settings: 6 general medical wards at Siriraj Hospital, Bangkok, Thailand

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients
* Received at least one dose of controlled antibiotics (Piperacillin/Tazobactam, Imipenem/Cilastatin, Meropenem or Doripenem)
* Each patient may be enrolled more than once, if he/she receives the controlled antibiotic for a new episode of infection (at least 48 hour apart)

Exclusion Criteria:

* Died prior to receive the controlled antibiotic

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 984 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Defined Daily Dose (DDD) of antibiotics | Participants will be followed for the total duration of antibiotic therapy for that given infection, an expected average of 2 weeks
  DDD of antibiotic use for that given infection (all antibiotics and controlled antibiotics)

SECONDARY OUTCOMES:
Total duration of antibiotic use | Participants will be followed for the total duration of antibiotic therapy for that given infection, an expected average of 2 weeks
  Total duration of antibiotic use for that given infection (all antibiotics and controlled antibiotics)

OTHER OUTCOMES:
Clinical response | at the end of therapy and at discharge (an average duration of antibiotic therapy is 2 weeks, an average length of stay is 3 weeks)
  Clinial response (cure, improved, not improved, dead and refer) at the end of therapy and at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Pinyo Rattanaumpawan, MD, MSCE, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Rattanaumpawan P, Upapan P, Thamlikitkul V. A noninferiority cluster-randomized controlled trial on antibiotic postprescription review and authorization by trained general pharmacists and infectious disease clinical fellows. Infect Control Hosp Epidemiol. 2018 Oct;39(10):1154-1162. doi: 10.1017/ice.2018.198. Epub 2018 Aug 29. PMID 30156171